CLINICAL TRIAL: NCT01293851
Title: Characterization of the Molecular-Genetic Mechanisms Associated With Chemotherapy-Induced Peripheral Neuropathy Progression
Brief Title: Molecular-Genetic Mechanisms Associated With Chemotherapy-Induced Nerve Damage
Status: Terminated | Type: Observational
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110065; 11-NR-0065
Record Dates: First submitted 2011-01-25; First posted 2011-02-11 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2012-11-13

CONDITIONS: Peripheral Neuropathic Pain; Neurotoxicity; Cancer
Keywords: Biomarkers; Gene Expression; Neuropathic Pain; Neurotoxicity; Chemotherapy; Peripheral Neuropathic Pain; Cancer
MeSH Terms: conditions — Neurotoxicity Syndromes; Neoplasms; Neuralgia

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Docetaxel, the most commonly used drug for the treatment of invasive breast cancer, has been shown to prolong the lives of women with breast cancer and prevent the cancer from spreading or returning. However, docetaxel is known to cause nerve damage, including numbness, tingling, and pain, in 50 to 90 percent of breast cancer patients. This nerve damage is called peripheral neuropathy, and can be so severe that treatment with docetaxel may need to be stopped. Researchers are interested in studying docetaxel-related nerve damage to determine whether certain genetic factors may predispose women to developing this condition, and to more closely investigate the specific effects of docetaxel on the nervous system

Objectives:

- To examine nerve damage in women with breast cancer who are being treated with docetaxel.

Eligibility:

- Women at least 18 years of age who have been diagnosed with invasive breast cancer and are scheduled to have docetaxel treatment.

Design:

* Participants will be screened with a full medical history and physical examination, as well as blood and urine tests and imaging studies.
* This study requires seven visits, one before the start of chemotherapy and six after the scheduled treatment visits. Study procedures at each visit will take 30 to 45 minutes and will be done in parallel with scheduled chemotherapy visits.
* At the first visit, participants will provide blood samples; complete questionnaires to rate and describe any existing pain, numbness, or tingling in hands and feet before the start of chemotherapy; have nerve conduction tests; and have a skin biopsy.
* At each visit following docetaxel treatment, participants will complete questionnaires to rate and describe any pain, numbness, or tingling during the course of chemotherapy. Participants will provide blood samples at every visit and have nerve conduction tests during the second, fourth, and sixth visits. Participants will also have a second skin biopsy, either from a site that appears to be experiencing nerve damage or (for those who are not developing nerve damage symptoms) from a site near the first biopsy location.

DETAILED DESCRIPTION:
Objective: Chemotherapy-induced peripheral neuropathy (CIPN) is one of the most debilitating side effects of neurotoxic chemotherapy, and can significantly interfere with patient quality of life (QOL) and the administration of antineoplastic therapy. There is no currently approved safe and effective treatment for CIPN. This protocol will explore the molecular-genetic mechanisms associated with the natural history of CIPN progression by (1) identification of differentially expressed genes and proteins as biomarkers for the onset of CIPN; (2) evaluation of the relationship between biomarkers and the severity of CIPN during the observation period, and (3) determining the relationship between molecular-genetic biomarkers, morphological changes in small nerve fiber and the severity of neuropathic symptoms.

Study population: Cancer patients who plan to receive chemotherapy treatment with either taxane class, vinca alkaloid class, platinum compounds or bortezomib.

Design: This is a prospective, exploratory, natural history study to identify the molecular-genetic mechanisms involved in chemotherapy-induced neuropathy in cancer patients. A physician-based neuropathy scale, patient neurotoxocity questionnaire, and the total neuropathy score will be used to measure the severity of peripheral neuropathy at baseline and after completion of each cycle of chemotherapy infusion. Whole peripheral blood and skin biopsy (only from patients who consent to biopsies) will be collected at baseline and after a subsequent infusion cycle to evaluate gene/protein expression and immunohistochemical labeling at peripheral sites of neuropathic injury. Microarray gene expression analysis will be employed to identify differential regulation of genes involved in the development of CIPN at the different time points compared with gene expression from the baseline samples. Genes of interest will be validated by qRT-PCR to identify novel pharmacological targets to be evaluated in future prospective studies. Protein levels corresponding to the changes in gene expression will be evaluated using ELISA and verified by Western blotting.

Outcome measures: The primary outcome of the study will be the changes in gene and protein expression in the peripheral blood and skin biopsy among cancer patients undergoing chemotherapy. The secondary outcome will be the relationship between the molecular-genetic biomarkers identified and the presence of peripheral neuropathic symptoms and their impacts on patient s QOL.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must meet all of the following to be eligible for enrollment:

* Age: 18 years and older
* Both male and female cancer patients will be recruited in this study. However, data will be separately assessed between males and females due to the differences in incidence, etiology and hormonal dependence which may confound the final data analyses.
* Ability to provide informed consent
* Cancer patients scheduled to undergo chemotherapy with taxane class, vinca alkaloid class, platinum compounds or bortezomib

EXCLUSION CRITERIA:

* Patients with any one of the following will be excluded:
* Unable to provide their own informed consent
* Have had prior radiotherapy
* Pre-existing documented neuropathy or risk factors for neuropathy that may confound the analysis of factors associated with CIPN such as:
* Diabetes mellitus
* Uremia
* Vitamin B12 deficiency
* Peripheral vascular disease
* Documented Thyroid dysfunction with on-going treatment. The patients who have thyroid dysfunction may also manifest the peripheral neuropathic symptoms such as numbness and tingling on their feet and hands. The medications used to treat hypothyroidism may confound the study data assessment.
* Previous history of alcoholism (beriberi) or drug abuse
* Rheumatoid arthritis
* Lupus
* Amyloidosis
* Sarcoidosis
* Other drug-induced neuropathy that may confound the analysis associated with CIPN such as:
* Thalidomide
* Isoniazid
* Trichloroethylene
* Hydralazine
* Disulfiram
* Nitrofurantoin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-12-22; Study Completion 2012-11-13

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Min Wang, M.D., Principal Investigator — National Institute of Nursing Research (NINR)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hoyert DL, Heron MP, Murphy SL, Kung HC. Deaths: final data for 2003. Natl Vital Stat Rep. 2006 Apr 19;54(13):1-120. PMID 16689256
- [Background] Thase ME, Frank E, Mallinger AG, Hamer T, Kupfer DJ. Treatment of imipramine-resistant recurrent depression, III: Efficacy of monoamine oxidase inhibitors. J Clin Psychiatry. 1992 Jan;53(1):5-11. PMID 1737741
- [Background] Cmelak AJ, Murphy BA, Burkey B, Douglas S, Shyr Y, Netterville J. Taxane-based chemoirradiation for organ preservation with locally advanced head and neck cancer: results of a phase II multi-institutional trial. Head Neck. 2007 Apr;29(4):315-24. doi: 10.1002/hed.20522. PMID 17252600